CLINICAL TRIAL: NCT04913194
Title: A Pilot Trial of A Two-Session Exposure Treatment and Parent Training for Picky Eating Consistent With an Avoidant-Restrictive Food Intake Disorder (ARFID) Diagnosis
Brief Title: A Two-Session Exposure Treatment and Parent Training for ARFID
Acronym: ARFID-PTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University at Albany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21E001
Record Dates: First submitted 2021-04-12; First posted 2021-06-04 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Avoidant Restrictive Food Intake Disorder
Keywords: Parent training; Exposure; ARFID; Picky eating; Brief intervention; Virtual intervention
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Food Fussiness

STUDY DESIGN:
Intervention Model Description: Two-arm waitlist control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants in this arm will receive the intervention within 2 weeks of completing the intake session.
  Interventions: Behavioral: ARFID-PTP
- Waitlist Control (Other): Participants in this arm will not receive any intervention for two weeks. Participants will complete the treatment after 4-6 weeks of being on the waitlist after their intake session.
  Interventions: Behavioral: ARFID-PTP

INTERVENTIONS:
Behavioral: ARFID-PTP — ARFID-PTP is a two-session virtual protocol using psychoeducation, parent training skills, and exposure to decrease picky eating symptoms consistent with an ARFID diagnosis.

SUMMARY:
This study aims to assess the acceptability, feasibility, and preliminary efficacy of a two-session, virtual parent-training exposure protocol for children ages 5-12 who experience picky eating consistent with an Avoidant-Restrictive Food Intake Disorder (ARFID) diagnosis.

DETAILED DESCRIPTION:
Potential subjects aged 5 to 12 years with picky eating symptoms consistent with an ARFID diagnosis, as determined by the Pica, ARFID, Rumination Disorder Interview, a semi-structured diagnostic interview, will be recruited via social media and local doctor's offices. Eligible subjects will complete informed consent and an intake session. Participants will then be randomized to an immediate treatment group, in which they will begin treatment the following week, or a 4-week waitlist condition, in which they will wait four weeks to begin treatment. All participants will have the opportunity to receive the treatment, ARFID Parent Training Program or "ARFID-PTP." ARFID-PTP was adapted from a seven-session parent-training for extremely picky eating behaviors to examine the efficacy of a two-session, virtual protocol on increasing food intake and decreasing selective eating. The two virtual treatment sessions will include psychoeducation, parent-training skills, and exposure protocol. There will be 5 major assessment time points: intake, end of treatment, 4-weeks post-treatment, 3-months post-treatment, and 6-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 5-12
* Child meets criteria for ARFID using the Pica, ARFID, Rumination Disorder Interview
* Established care with a primary care provider
* Not engaging in other medication or psychotherapy for ARFID during this treatment trial
* Fluently speak and read English

Exclusion Criteria:

* Child or parent experiencing suicidal thoughts
* Child or parent experiencing psychotic symptoms
* Child has a cognitive functioning disability

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | Enrollment
  Recruitment rates will be measured by the average number of participants recruited each month.
Retention Feasibility | Through study completion, up to 9 months
  Retention rates will be measured as the percentage of families who begin treatment and complete all follow-up time points.
Acceptability of exposure protocol | Through study completion, up to 9 months
  Acceptability of exposure will be measured as a percentage of number of daily food exposures the family completes at all follow-up time points.
Credibility of treatment | After week 2 of treatment
  The Credibility and Expectancy Questionnaire is a 6-item measure of treatment credibility and how much participants think and feel treatment will work.
Acceptability of treatment | After week 2 of treatment
  Parents will self-report the acceptability of treatment by selecting the extent to which they agree with statements such as "I would refer this treatment to a friend" or "I am satisfied with this treatment."
Acceptability of treatment at 1-month follow-up | 1 month
  Parents will self-report the acceptability of treatment by selecting the extent to which they agree with statements such as "I would refer this treatment to a friend" or "I am satisfied with this treatment."

SECONDARY OUTCOMES:
Pica, ARFID, Rumination Disorder Interview (PARDI) | Change between intake and 3-month follow-up
  The PARDI is a semi-structured interview assessing for diagnostic criteria of ARFID, as well as subtype classification and severity ratings. Parents will be assessed using the PARDI.
Treatment Efficacy: Foods in Regular Rotation | Through study completion, up to 9 months
  Parents will self-report the number of new foods a child has included in "regular rotation" i.e., is able to eat a full serving size regularly.
Behavioral Pediatric Feeding Assessment Scale | Through study completion, up to 9 months
  The Behavioral Pediatric Feeding Assessment Scale is a well-validated measure of child's eating behaviors and parental perception of eating behaviors.
Treatment Efficacy: Goal Progress | Through study completion, up to 9 months
  Treatment goals will be assessed using the ARFID-specific treatment goal checklist established by Bryant-Waugh in 2020 via the Maudsley Centre for Child and Adolescent Eating Disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney E Breiner, MA, Principal Investigator — University at Albany, State University of New York
Locations (1):
- University at Albany, State University of New York, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breiner CE, Miller ML, Hormes JM. ARFID Parent Training Protocol ("ARFID-PTP"): Results of a Randomized Pilot Trial Evaluating a Brief, Parent-Training Program for Avoidant/Restrictive Food Intake Disorder. Int J Eat Disord. 2024 Nov;57(11):2306-2317. doi: 10.1002/eat.24269. Epub 2024 Jul 19. PMID 39031449